CLINICAL TRIAL: NCT03542981
Title: Is Interferential Current Effective in the Management of Pain, Range of Motion, Edema Following Total Knee Arthroplasty Surgery?: Randomized Double-blind Controlled Trial
Brief Title: Interferential Current Therapy After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Resul KADI, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TKP35IF
Record Dates: First submitted 2018-05-07; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Total Knee Arthroplasty
Keywords: pain; surgery; interferential current; total knee arthroplasty
MeSH Terms: conditions — Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferential Current Treatment (Active Comparator): Interferential Current group received interferential current treatment 30 minutes, 2 times a day for 5 days after the surgery.
  Interventions: Device: Interferential Current
- Sham Interferential Current Treatment (Sham Comparator): In the sham interferential Current treatment, no electrical stimulation was applied to the probes with the same pads for the same time.
  Interventions: Device: Sham Interferential Current

INTERVENTIONS:
Device: Interferential Current
  Arms: Interferential Current Treatment
Device: Sham Interferential Current
  Arms: Sham Interferential Current Treatment

SUMMARY:
Interferential current is widely used as a popular treatment in painful musculoskeletal disorders. And total knee arthroplasty patients present with extreme pain immediately after surgery. So this study is aimed to investigate the effectiveness of interferential current implementation following total knee arthroplasty surgery. In this study interferential current compared with sham interferential current . Patients were assessed with pain, range of motion , edema and the amount of used paracetamol.

DETAILED DESCRIPTION:
A total of 132 patients ranging in 60-85 years who were undergoing their first total knee arthroplasty due to knee OA were recruited into a randomized, double-blind, prospective and controlled study. Participants were recruited at the Orthopedics and Traumatology inpatient clinic. The patients were seen postoperative first day and were assigned to receive either interferential current or sham interferential current by block randomization. After the procedure was explained to each subject, interferential current treatment was applied 2 times for 5 days, each treatment was continued approximately 30 minutes. Four electrodes were used to deliver quadripolar interferential current Subjects were told that in order to produce an effect, the intensity of the stimulator must be maintained at a "strong but comfortable level" at all times. The sham interferential current treatment consisted of the placement of the same pads for the same time but no electrical stimulation was applied to the probes. At the same time, all patients received standard postoperatively rehabilitation program. Patients were assessed with pain, range of motion , edema and the amount of used paracetamol.

ELIGIBILITY:
Inclusion Criteria:

•Patients who underwent total knee arthroplasty surgery

Exclusion Criteria:

* Patients who had experienced of any electrotherapy prior to the TKA to be sure blinding of therapy
* Patients who had history of any contraindication for electrotherapy
* Patients who had chronic pain rather than knee OA
* Patients who had experienced a known or suspected joint infection or a specific condition (ie, peripheral or central nervous system lesions, neoplasm, diabetes mellitus, osteonecrosis, recent trauma and pacemaker)
* Patients who had history of stroke, central nervous disease, mental impairment or poor general health status that would interfere with functional assessments during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-09-09 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain from baseline measured by visual analog scale | Change in pain measured 5th and 30th days after surgery
  Pain intensity that was measured by visual analog scale (minimum score:0; maximum score:100)(higher values represent worse outcome)

SECONDARY OUTCOMES:
Change of Range of Motion from baseline | Change of Range of Motion measured 5th and 30th days after surgery
  The measurement of the range of the motion was performed by a goniometer of active extension and flexion (higher values represent better outcome)
Change of Edema from baseline | Change of Edema measured 5th and 30th days after surgery
  Edema as a change in circumference from the preoperative value was measured by a meter (higher values represent worse outcome)
Amount of used paracetamol | 5th and 30th days after surgery
  the paracetamol intake was recorded as gr. (higher values represent worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: mehmet r kadı, MD, Principal Investigator — Ege University School of Medicine; Simin Hepguler, prof, Study Director — Ege University School of Medicine; Funda C Atamaz, prof, Study Chair — Ege University School of Medicine; Emine Dede, md, Study Chair — Ege University School of Medicine; Semih Aydogu, prof, Study Chair — Ege University School of Medicine; Kemal Aktuğlu, prof, Study Chair — Ege University School of Medicine; Nadir Ozkayın, prof, Study Chair — Ege University School of Medicine; Cihat Ozturk, prof, Study Chair — Ege University School of Medicine
Locations (1):
- Ege University School of Medicine Hospital, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No